CLINICAL TRIAL: NCT00424008
Title: A 52-Week Efficacy and Safety Non-Inferiority Study of Fluticasone Propionate/Salmeterol 250/50mcg BID Delivered by Dry Powder Inhaler (Diskus) Versus Mometasone Furoate/Formoterol Fumarate 200/10mcg BID Delivered by Pressurized Metered-Dose Inhaler in Persistent Asthmatics Previously Treated With Medium Doses of Inhaled Glucocorticosteroids
Brief Title: Study of Inhaled Glucocorticosteroids/Long-Acting Bronchodilator Drugs in Subjects With Asthma That Have Been Taking Inhaled Glucocorticosteroids (Study P04705AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P04705; SCH 418131
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: Glucocorticosteroids; Dry Powder Inhaler; Bronchodilator; Metered-Dose Inhaler
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Formoterol Fumarate; Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MF/F MDI 200/10 mcg BID (Experimental): Mometasone furoate 200 mcg and formoterol 10 mcg fixed dose combination taken twice daily.
  Interventions: Drug: Mometasone furoate/formoterol (MF/F) MDI
- F/SC DPI 250/50 mcg BID (Active Comparator): Fluticasone propionate/salmeterol (F/SC) 250/50 mcg BID
  Interventions: Drug: Fluticasone propionate/salmeterol (F/SC) DPI

INTERVENTIONS:
Drug: Mometasone furoate/formoterol (MF/F) MDI — MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 52 weeks.
  Other Names: SCH 418131
  Arms: MF/F MDI 200/10 mcg BID
Drug: Fluticasone propionate/salmeterol (F/SC) DPI — Fluticasone propionate 250 mcg and salmeterol 50 mcg fixed dose combination dry powder inhaler taken twice daily for 52 weeks.
  Other Names: Advair Diskus in the US/Seretide Diskus outside the US
  Arms: F/SC DPI 250/50 mcg BID

SUMMARY:
This study is being conducted to demonstrate the non-inferiority between two inhaled glucocorticosteroids and long-acting bronchodilator combination drugs called mometasone furoate/formoterol fumarate in a metered-dose inhaler (MDI) and fluticasone propionate/salmeterol in a dry powder inhaler (DPI) on lung function. Information on the onset of action, the overall safety, and how the drugs control asthma will also be assessed. The study is approximately 1 year in duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of asthma for at least 12 months' duration.
* A participant must have been using a medium daily dose of inhaled glucocorticosteroids (alone or in combination with long-acting beta 2-agonist [LABA]) for at least 12 weeks and must have been on a stable regimen for at least 2 weeks prior to Screening.
* If there is no inherent harm in changing the participant's current asthma therapy, the participant must be willing to discontinue his/her prescribed inhaled glucocorticosteroid (ICS) or ICS/LABA prior to initiating MF MDI run-in medication.
* The diagnosis of asthma must be documented by either demonstrating an increase in absolute forced expiratory volume in 1 second (FEV1) of at least 12% and a volume increase of at least 200 mL within approximately 15 to 20 minutes after administration of 4 inhalations of albuterol/salbutamol or of nebulized short-acting beta 2-agonist (SABA) OR peak expiratory flow (PEF) variability of more than 20% OR a diurnal variation PEF of more than 20% based on the difference between pre-bronchodilator (before taking albuterol/salbutamol) morning value and the post-bronchodilator value (after taking albuterol/salbutamol) from the evening before, expressed as a percentage of the mean daily PEF value on any day during the open-label Run-in Period.
* A participant must have a history of >= 2 asthma-related unscheduled visits to a physician or to an emergency room within the past year AND >= 3 asthma-related unscheduled visits within the past 2 years.
* Prior to randomization participants must have used a total of 12 or more inhalations of SABA rescue medication during the last 10 days of run-in.
* Clinical laboratory tests (complete blood counts [CBC], blood chemistries, including serum pregnancy for females of child-bearing potential, and urinalysis) conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor before the participant is instructed to start using open-label MF MDI run-in medication.
* An electrocardiogram (ECG) performed at the Screening Visit, using a centralized trans-telephonic technology, must be clinically acceptable to the investigator.
* A chest x-ray performed at the Screening Visit, or within 12 months prior to the Screening Visit, must be clinically acceptable to the investigator.
* A non-pregnant female participant of childbearing potential must be using a medically acceptable, adequate form of birth control. A female participant of childbearing potential must have a negative serum pregnancy test at Screening in order to be considered eligible for enrollment.

Exclusion Criteria:

* A participant who demonstrates a change in absolute FEV1 of > 20% at any time between the Screening and Baseline Visits on any 2 consecutive days between the Screening and Baseline visits.
* A participant who requires the use of greater than 8 inhalations per day of SABA MDI or 2 or more nebulized treatments per day of 2.5 mg SABA on any 2 consecutive days between the Screening and Baseline Visits.
* A participant who experiences a decrease in AM or PM PEF below the Run-in Period stability limit on any 2 consecutive days prior to randomization. The average AM and average PM PEF respective values from the preceding 7 days are added, divided by the number of non-missing values, and multiplied by 0.70 to determine the stability limit.
* A participant who experiences a clinical asthma exacerbation: defined as a clinical deterioration of asthma as judged by the clinical investigator between the Screening and Baseline Visits, that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication (including oral or other systemic corticosteroids, but allowing SABA).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernstein DI, Hebert J, Cheema A, Murphy KR, Cherrez-Ojeda I, Matiz-Bueno CE, Kuo WL, Nolte H. Efficacy and onset of action of mometasone furoate/formoterol and fluticasone propionate/salmeterol combination treatment in subjects with persistent asthma. Allergy Asthma Clin Immunol. 2011 Dec 7;7(1):21. doi: 10.1186/1710-1492-7-21. PMID 22152089
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to standardize treatment prior to randomization, participants entered a 2- to 4-week open-label Run-in period where they received MF MDI 200 mcg BID. Participants who continued to meet eligibility criteria at the completion of the Run-in Period were randomized into the study.
Groups:
- MF/F MDI 200/10 mcg BID: Mometasone furoate 200 mcg and formoterol 10 mcg (MF/F) fixed dose combination taken twice daily (BID) via a metered-dose inhaler (MDI).
- F/SC DPI 250/50 mcg BID: Fluticasone propionate/salmeterol (F/SC) 250/50 mcg Dry Powder Inhaler (DPI) BID
Period: Overall Study
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID
Started | 371 | 351
Completed | 22 | 16
Not Completed | 349 | 335
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 40 | 34
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Noncompliance with protocol | 13 | 7
Not completed — Did not meet protocol eligibility | 16 | 21
Not completed — Administrative | 266 | 257

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID | Total
Number analyzed (Participants) | 371 | 351 | 722
Age, Customized [Number; unit: participants]
  12 to <18 years | 22 | 18 | 40
  18 to <65 years | 321 | 308 | 629
  >=65 years | 28 | 25 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 220 | 459
  Male | 132 | 131 | 263

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Curve From 0 to 12 Hours [AUC](0-12 hr) of the Change From Baseline to the Week 12 Endpoint in Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline to Week 12
Population: Efficacy analyses were based on randomized subjects with Baseline and any post-baseline data (intent-to-treat principle). The standard deviation is pooled. Least Squares Mean scores are obtained from an analysis of covariance model correcting for treatment, site effects, and the Baseline FEV1 (liters) as a covariate.
Measure: Least Squares Mean (Standard Deviation); unit: Liter x hour
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID
Number analyzed (Participants) | 366 | 346
Liter x hour | 3.43 (3.83) [-0.56 to 0.79] | 3.24 (3.83) [-0.56 to 0.79]

2. Secondary Outcome: Onset-of-action Based on Change From Baseline FEV1 at the 5 Min Pulmonary Function Test (PFT) Assessment on Day 1
Description: PFTs, including FEV1, were done on Day 1. Evaluations included 30 min before and immediately before the first dose, the mean of which was Baseline, and at intervals from 5 min to 12 hrs postdose. Onset of action was defined as statistically significant improvement of MF/F over F/SC in Change from Baseline FEV1 at the 5-min postdose evaluation on Day 1. The same series of PFTs were done at Week 12. Change from Baseline to Week 12 evaluations were calculated using the same Day 1 predose scores for Baseline. The Week-12 evaluation consisted of AUC FEV1 scores across the 12-hour postdose interval.
Time Frame: Baseline to 5 minutes post-dose on Day 1
Population: Participants with data at Day One 5 minutes post-dose.
  The standard deviation is pooled. Least Squares Mean scores are obtained from an analysis of covariance model correcting for treatment, site effects, and the Baseline FEV1 (liters) as a covariate.
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID
Number analyzed (Participants) | 365 | 348
Liters | 0.20 (0.20) | 0.09 (0.20)

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Total Score at Week 12 Endpoint
Description: The Asthma Control Questionnaire (ACQ) by Juniper et al. is a mean of 7 equally weighted composite scores; each scaled from 0=best case scenario to 6=worst case scenario on an integer scale. Composites include the following: How Often Woken by Asthma, How Bad Were Asthma Symptoms When You Woke, Activity Limitations, Shortness of Breath, Wheezing, Average Daily Short-Acting Beta 2-Agonist (SABA) Puffs, and physician-evaluated lung function. With the exception of physician-evaluated lung function collected at the visit, evaluations were over the last week recall period.
Time Frame: Baseline to Week 12
Population: Efficacy analyses were based on randomized subjects with Baseline and any postbaseline data (intent-to-treat principle).
  The standard deviation is pooled. Least Squares Mean scores are obtained from an analysis of covariance model correcting for treatment, site effects, and the Baseline ACQ score as a covariate.
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID
Number analyzed (Participants) | 350 | 331
Scores on a scale | -0.65 (0.61) | -0.65 (0.61)

4. Secondary Outcome: The Proportion of Symptom-free Days and Nights (Combined) Over the 12-week Treatment Period.
Description: For each day of the evaluation period, symptoms were collected in the morning for the night's evaluation, and in the evening for the day's evaluation. Symptoms included coughing, wheezing, and difficulty breathing, each integer-scaled from 0=none to 3=severe. A symptom-free Day/Night is defined as a combined score of 0 across the morning and evening evaluations. The proportion of 0 scores across the Baseline period, and across the 12-week treatment period, is calculated to determine the overall proportion of symptom-free Days/Nights for each of these periods.
Time Frame: Baseline to Week 12
Population: Efficacy analyses were based on randomized subjects with Baseline and any post-baseline data (intent-to-treat principle).
  The standard deviation is pooled. Least Squares Mean scores are obtained from an analysis of covariance model correcting for treatment, site effects, and the Baseline proportion of symptom-free days/nights as a covariate.
Measure: Least Squares Mean (Standard Deviation); unit: Proportion of symptom-free days/nights
Arm/Group | MF/F MDI 200/10 mcg BID | F/SC DPI 250/50 mcg BID
Number analyzed (Participants) | 364 | 349
Proportion of symptom-free days/nights
  Baseline (over the last week prior to first dose) | 0.19 (0.28) | 0.18 (0.28)
  Actual proportion over the 12-wk treatment period | 0.42 (0.32) | 0.43 (0.32)
  Change from Baseline to over the 12-wk tx period | 0.24 (0.32) | 0.25 (0.32)

ADVERSE EVENTS:
Description: This study included a 2 to 4-week open-label (OL) run-in period prior to randomization. The OL MF MDI 200 mcg BID group includes all screened participants who were administered at least one dose. Participants who continued to meet eligibility criteria at the completion of the OL run-in period were subsequently randomized to either MF/F or F/SC.
Groups:
- Open-label (OL) MF MDI * 200 MCG BID: Mometasone furoate 200 mcg taken twice daily (BID) via a metered-dose inhaler (MDI).
- MF/F MDI * 200/10 MCG * BID: Mometasone furoate 200 mcg and formoterol 10 mcg (MF/F) fixed dose combination taken twice daily (BID) via a metered-dose inhaler (MDI).
- F/SC DPI * 250/50 MCG BID: Fluticasone propionate/salmeterol (F/SC) 250/50 mcg Dry Powder Inhaler (DPI) BID
Arm/Group | Open-label (OL) MF MDI * 200 MCG BID | MF/F MDI * 200/10 MCG * BID | F/SC DPI * 250/50 MCG BID
Serious Adverse Events (participants affected / at risk) | 0/983 | 6/371 | 8/351
Other Adverse Events (participants affected / at risk) | 43/983 | 85/371 | 77/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (OL) MF MDI * 200 MCG BID (N=983) | MF/F MDI * 200/10 MCG * BID (N=371) | F/SC DPI * 250/50 MCG BID (N=351)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (OL) MF MDI * 200 MCG BID (N=983) | MF/F MDI * 200/10 MCG * BID (N=371) | F/SC DPI * 250/50 MCG BID (N=351)
Nasopharyngitis (Infections and infestations) | 5 (5) | 33 (38) | 24 (27)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 25 (31) | 16 (20)
Headache (Nervous system disorders) | 37 (50) | 42 (109) | 45 (88)

LIMITATIONS AND CAVEATS:
The sponsor closed the study early, at 12 weeks treatment, for reasons that were not safety related. No efficacy analysis of data collected beyond 12 weeks of treatment was performed. All safety data were examined regardless of treatment duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results without prior sponsor written consent. The investigator agrees to provide to the sponsor, 45 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues/disagreement.